CLINICAL TRIAL: NCT01603459
Title: Prospective, Open-label, Non-randomized, Single-arm, Multi-center Dose Titration Study to Investigate the Safety and Efficacy of NT 201 in Subjects Deemed to Require Total Body Doses of 800 U of NT 201 During the Course of the Study for the Treatment of Upper and Lower Limb Spasticity of the Same Body Side Due to Cerebral Causes
Brief Title: Efficacy and Safety Dose Titration Study of Botulinum Toxin Type A to Treat Spasticity in the Leg and Arm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ60201_3053_1; 2010-020886-26 (EudraCT Number)
Record Dates: First submitted 2012-04-17; First posted 2012-05-22 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Spasticity of the Upper and Lower Limb Due to Cerebral Causes
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IncobotulinumtoxinA (Xeomin) (up to 800 Units) (Experimental): IncobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection
  Interventions: Drug: IncobotulinumtoxinA

INTERVENTIONS:
Drug: IncobotulinumtoxinA — Subjects to receive up to 3 injection cycle, with the dose titrated from 400 units to up to 800 units.
  For each injection session: solution prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 400-800 units, volume 2.0 mL per 100 units; Mode of administration: intramuscular injection.

SUMMARY:
The purpose of this study is to determine whether injections with increasing doses (up to 800 units) of Botulinum toxin type A into muscles of the leg and/or arm are safe and effective in treating patients with spasticity on one body side due to cerebral causes.

DETAILED DESCRIPTION:
A dose-titration approach will be used over three injection cycles, with a flexible observation period after injections of 12-16 weeks and a total duration of up to 48 weeks. Cycle 1 and 2: upper and/or lower limb to be treated; Cycle 3: upper and lower limb to be treated.

ELIGIBILITY:
Inclusion Criteria:

* Upper and lower limb spasticity of the same body side due to cerebral causes
* Time since event leading to spasticity in the target body side greater than 12 weeks
* Need for 800 units Botulinum toxin type A

Exclusion Criteria:

* Body weight below 50kg
* Fixed contractures of the target joint
* Generalized disorders of muscle activity like Myasthenia gravis that preclude use of Botulinum toxin type A
* Infection at the injection site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals
Locations (33):
- United States (6):
  - Merz Investigational Site # 001197, Doral, Florida
  - Merz Investigational Site # 001235, Indianapolis, Indiana
  - Merz Investigational Site # 001191, New York, New York
  - Merz Investigational Site #001238, Charlotte, North Carolina
  - Merz Investigational Site # 001232, Cleveland, Ohio
  - Merz Investigational Site #001237, Milwaukee, Wisconsin
- Canada (2):
  - Merz Investigational Site # 001203, Calgary, AB
  - Merz Investigational site #001195, Edmonton, AB
- France (3):
  - Merz Investigational Site # 033018, Garches
  - Merz Investigational Site #033049, Montpellier
  - Merz Investigational Site # 033050, Nîmes
- Germany (8):
  - Merz Investigational Site #049191, Aachen
  - Merz Investigational Site #049297, Bad Aibling
  - Merz Investigational Site #049022, Beelitz-Heilstätten
  - Merz Investigational Site #049298, Berlin
  - Merz Investigational Site # 049153, Giessen
  - Merz Investigational Site #049295, Göttingen
  - Merz Investigational Site #049300, Nümbrecht
  - Merz Investigational Site #049296, Tübingen
- Italy (7):
  - Merz Investigational Site # 039005, Lecco
  - Merz Investigational Site # 039010, Milan
  - Merz Investigational Site # 039015, Milan
  - Merz Investigational Site # 039017, Novara
  - Merz Investigational Site #039013, Passignano sul Trasimeno
  - Merz Investigational Site #039016, San Giovanni Rotondo
  - Merz Investigational Site #039014, Verona
- Merz Investigational Site #047001, Bergen, Norway
- Portugal (2):
  - Merz Investigational Site # 351003, Lisbon
  - Merz Investigational Site # 351001, Lisbon
- Spain (4):
  - Merz Investigational Site #034007, Madrid
  - Merz Investigational Site #034022, Manresa
  - Merz Investigational Site #034025, Málaga
  - Merz Investigational Site #034024, Santander

REFERENCES:
- [Result] Wissel J, Bensmail D, Ferreira JJ, Molteni F, Satkunam L, Moraleda S, Rekand T, McGuire J, Scheschonka A, Flatau-Baque B, Simon O, Rochford ET, Dressler D, Simpson DM; TOWER study investigators. Safety and efficacy of incobotulinumtoxinA doses up to 800 U in limb spasticity: The TOWER study. Neurology. 2017 Apr 4;88(14):1321-1328. doi: 10.1212/WNL.0000000000003789. Epub 2017 Mar 10. PMID 28283596
- [Derived] Fheodoroff K, Scheschonka A, Wissel J. Goal analysis in patients with limb spasticity treated with incobotulinumtoxinA in the TOWER study. Disabil Rehabil. 2022 Apr;44(8):1367-1373. doi: 10.1080/09638288.2020.1804627. Epub 2020 Aug 17. PMID 32805151
- [Derived] Fheodoroff K, Rekand T, Medeiros L, Kossmehl P, Wissel J, Bensmail D, Scheschonka A, Flatau-Baque B, Simon O, Dressler D, Simpson DM. Quality of life in subjects with upper- and lower-limb spasticity treated with incobotulinumtoxinA. Health Qual Life Outcomes. 2020 Mar 4;18(1):51. doi: 10.1186/s12955-020-01304-4. PMID 32131842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical study was conducted at 30 sites located in Canada, France, Germany, Italy, Norway, Portugal, Spain, and the United States of America.
Groups:
- IncobotulinumtoxinA (Xeomin) (up to 800 Units): IncobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection.
  IncobotulinumtoxinA: Subjects to receive up to 3 injection cycle, with the dose titrated from 400 units to up to 800 units.
  For each injection session: solution prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 400-800 units, volume 2.0 mL per 100 units; Mode of administration: Intramuscular injection.
Period: Overall Study
Arm/Group | IncobotulinumtoxinA (Xeomin) (up to 800 Units)
Started | 155
Completed | 137
Not Completed | 18
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 3
Not completed — Predefined discontinuation criteria | 3
Not completed — Non-compliance | 1
Not completed — Administrative reason | 1

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) is the subset of all subjects who were exposed to study medication at least once.
Arm/Group | IncobotulinumtoxinA (Xeomin) (up to 800 Units)
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 104

OUTCOME MEASURES:

1. Secondary Outcome: Ashworth Scale (AS) Scores of the Target Joint Selected at Study Baseline Visit
Description: The AS is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: The full analysis set (FAS) is the subset of all subjects who were exposed to study medication at least once. Only subjects treated in the target joint in the respective cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit; IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1: Subjects to receive IncobotulinumtoxinA fixed total body dose of 400 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit; IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1: Subjects to receive IncobotulinumtoxinA fixed total body dose of 600 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit; IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1: Subjects to receive IncobotulinumtoxinA total body dose of 800 units Intramuscular injection.
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1
Number analyzed (Participants) | 154 | 154 | 151 | 148 | 140 | 138
units on a scale | 3.0 (0.7) | 2.1 (0.9) | 2.7 (0.7) | 2.0 (0.9) | 2.6 (0.8) | 1.7 (1.0)

2. Secondary Outcome: Change of Ashworth Scale (AS) Score of the Target Joint Selected at Study Baseline Visit From Injection Cycle Baseline Visits to Respective Control Visits
Description: as for outcome 1
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS), observed cases, only subjects treated in the target joint in the respective cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IncobotulinumtoxinA (Xeomin): Injection Cycle 1: Subjects to receive IncobotulinumtoxinA fixed total body dose of 400 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Injection Cycle 2: Subjects to receive IncobotulinumtoxinA fixed total body dose of 600 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Injection Cycle 3: Subjects to receive IncobotulinumtoxinA total body dose of 800 units Intramuscular injection.
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 154 | 148 | 138
units on a scale | -0.8 (0.9) | -0.8 (0.8) | -0.9 (0.9)

3. Secondary Outcome: Change of Ashworth Scale (AS) Score of the Target Joint Selected at Study Baseline Visit From Study Baseline Visit to Control Visits of Injection Cycles
Description: as for outcome 1
Time Frame: From Study Baseline to Week 4, 16-20 and 28-36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IncobotulinumtoxinA (Xeomin): Time Frame 1: Time frame 1 is from Study Baseline to Cycle 1 Control Visit. Subjects to receive IncobotulinumtoxinA fixed total body dose of 400 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Time Frame 2: Time frame 2 is from Study Baseline to Cycle 2 Control Visit. Subjects to receive IncobotulinumtoxinA fixed total body dose of 600 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Time Frame 3: Time frame 3 is from Study Baseline to Cycle 3 Control Visit. Subjects to receive IncobotulinumtoxinA total body dose of 800 units Intramuscular injection.
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 154 | 148 | 138
units on a scale | -0.8 (0.9) | -1.0 (0.9) | -1.3 (1.0)

4. Secondary Outcome: Change of Ashworth Scale (AS) Score of the Target Joint Selected at Study Baseline Visit From Study Baseline Visit to Injection Cycle Baseline Visits and End of Cycle 3 Visit
Description: as for outcome 1
Time Frame: From Study Baseline to Week 12-16, 24-32 and 36-48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IncobotulinumtoxinA (Xeomin): Timeframe 1: Time frame 1 is from Study Baseline to Cycle 2 Baseline. Subjects to receive IncobotulinumtoxinA fixed total body dose of 400 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Time Frame 2: Time frame 2 is from Study Baseline to Cycle 3 Baseline. Subjects to receive IncobotulinumtoxinA fixed total body dose of 600 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Time Frame 3: Time frame 3 is from Study Baseline to End of Cycle 3 Visit. Subjects to receive IncobotulinumtoxinA total body dose of 800 units Intramuscular injection.
Arm/Group | IncobotulinumtoxinA (Xeomin): Timeframe 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 151 | 140 | 137
units on a scale | -0.2 (0.7) | -0.3 (0.8) | -0.7 (0.9)

5. Secondary Outcome: Ashworth Scale (AS) Scores of Every Joint Affected by Clinical Patterns of Spasticity
Description: Clinical pattern treated at corresponding cycle of the same body side as the selected target joint. The AS is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective pattern in the respective injection cycle.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1
Number analyzed (Participants) | 155 | 155 | 152 | 152 | 140 | 140
units on a scale
  Internally rotated/extended/adducted shoulder: number analyzed (Participants) | 52 | 52 | 69 | 68 | 84 | 83
  Internally rotated/extended/adducted shoulder | 2.7 (0.6) | 2.2 (0.8) | 2.5 (0.8) | 2.0 (0.9) | 2.5 (0.8) | 1.9 (0.9)
  Flexed elbow: number analyzed (Participants) | 117 | 117 | 122 | 121 | 124 | 122
  Flexed elbow | 2.6 (0.7) | 1.9 (0.9) | 2.4 (0.7) | 1.7 (0.9) | 2.4 (0.8) | 1.4 (0.9)
  Extended elbow: number analyzed (Participants) | 11 | 11 | 16 | 15 | 19 | 19
  Extended elbow | 2.7 (0.5) | 1.8 (0.9) | 2.5 (0.6) | 2.1 (0.7) | 2.6 (0.6) | 1.7 (0.8)
  Pronated forearm: number analyzed (Participants) | 37 | 37 | 50 | 50 | 48 | 47
  Pronated forearm | 2.7 (0.7) | 1.6 (0.9) | 2.4 (0.8) | 1.7 (1.0) | 2.5 (0.7) | 1.4 (0.8)
  Flexed wrist: number analyzed (Participants) | 84 | 84 | 87 | 85 | 91 | 90
  Flexed wrist | 2.7 (0.8) | 1.8 (1.0) | 2.4 (0.9) | 1.5 (1.0) | 2.4 (0.8) | 1.4 (1.0)
  Clenched fist: number analyzed (Participants) | 96 | 96 | 110 | 108 | 110 | 108
  Clenched fist | 2.9 (0.7) | 2.0 (0.9) | 2.7 (0.8) | 1.8 (0.9) | 2.5 (0.7) | 1.5 (0.9)
  Thumb in palm: number analyzed (Participants) | 53 | 53 | 63 | 61 | 65 | 63
  Thumb in palm | 2.4 (0.9) | 1.5 (1.1) | 2.3 (0.9) | 1.4 (1.0) | 2.2 (0.8) | 1.3 (1.0)
  Flexed hip: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 5
  Flexed hip |  |  |  |  | 1.8 (0.8) | 1.4 (0.9)
  Adducted thigh: number analyzed (Participants) | 4 | 4 | 7 | 7 | 7 | 7
  Adducted thigh | 1.8 (0.5) | 1.5 (0.6) | 2.0 (1.2) | 1.9 (0.9) | 2.3 (0.8) | 2.0 (0.6)
  Internally rotated hip: number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 3
  Internally rotated hip | 3.0 (NA) — NA = data not available | 2.0 (NA) — NA = data not available | 2.0 (1.4) | 2.0 (1.4) | 2.7 (0.6) | 1.7 (0.6)
  Flexed knee: number analyzed (Participants) | 12 | 12 | 24 | 23 | 32 | 32
  Flexed knee | 2.4 (0.7) | 2.0 (0.7) | 2.4 (0.6) | 1.8 (0.7) | 2.5 (0.7) | 1.8 (1.0)
  Extended knee: number analyzed (Participants) | 11 | 11 | 22 | 21 | 27 | 26
  Extended knee | 2.6 (0.7) | 2.3 (0.9) | 2.1 (0.8) | 1.8 (0.9) | 2.2 (0.8) | 1.5 (0.8)
  Pes equinovarus: number analyzed (Participants) | 88 | 88 | 117 | 115 | 122 | 120
  Pes equinovarus | 2.8 (0.7) | 2.1 (0.9) | 2.6 (0.8) | 1.9 (1.0) | 2.5 (0.8) | 1.6 (0.9)
  Pes equinovalgus: number analyzed (Participants) | 5 | 5 | 10 | 10 | 8 | 8
  Pes equinovalgus | 2.8 (0.4) | 2.4 (1.3) | 2.6 (0.8) | 1.9 (0.7) | 2.3 (0.9) | 2.0 (1.1)
  Extended hallux: number analyzed (Participants) | 10 | 10 | 10 | 10 | 20 | 19
  Extended hallux | 1.7 (1.1) | 0.9 (0.7) | 1.8 (0.8) | 0.9 (0.7) | 1.9 (0.9) | 1.1 (0.8)
  Flexed toes: number analyzed (Participants) | 27 | 27 | 34 | 34 | 45 | 45
  Flexed toes | 1.8 (0.9) | 1.3 (0.8) | 1.6 (0.9) | 1.1 (0.8) | 1.9 (0.9) | 1.1 (0.8)

6. Secondary Outcome: Change of Ashworth Scale (AS) Score of Every Joint Affected by Clinical Patterns of Spasticity From Injection Cycle Baseline Visits to Respective Control Visits
Description: as for outcome 5
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective pattern of respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 155 | 152 | 140
units on a scale
  Internally rotated/extended/adducted shoulder: number analyzed (Participants) | 52 | 68 | 83
  Internally rotated/extended/adducted shoulder | -0.5 (0.8) | -0.6 (0.8) | -0.5 (0.8)
  Flexed elbow: number analyzed (Participants) | 117 | 121 | 122
  Flexed elbow | -0.7 (0.8) | -0.7 (0.8) | -0.9 (0.9)
  Extended elbow: number analyzed (Participants) | 11 | 15 | 19
  Extended elbow | -0.9 (0.8) | -0.5 (0.9) | -0.8 (0.8)
  Pronated forearm: number analyzed (Participants) | 37 | 50 | 47
  Pronated forearm | -1.1 (0.6) | -0.7 (0.7) | -1.0 (0.8)
  Flexed wrist: number analyzed (Participants) | 84 | 85 | 90
  Flexed wrist | -0.9 (0.8) | -0.9 (0.8) | -1.0 (0.9)
  Clenched fist: number analyzed (Participants) | 96 | 108 | 108
  Clenched fist | -0.9 (0.8) | -0.9 (0.8) | -1.1 (0.8)
  Thumb in palm: number analyzed (Participants) | 53 | 61 | 63
  Thumb in palm | -0.9 (1.0) | -0.9 (1.1) | -0.9 (1.0)
  Flexed hip: number analyzed (Participants) | 0 | 0 | 5
  Flexed hip |  |  | -0.4 (0.9)
  Aducted thigh: number analyzed (Participants) | 4 | 7 | 7
  Aducted thigh | -0.3 (0.5) | -0.1 (0.7) | -0.1 (1.0)
  Internally rotated hip: number analyzed (Participants) | 1 | 2 | 3
  Internally rotated hip | -1.0 (NA) — NA = data not available | 0.0 (0.0) | -1.0 (1.0)
  Flexed knee: number analyzed (Participants) | 12 | 23 | 32
  Flexed knee | -0.4 (0.5) | -0.6 (0.6) | -0.8 (0.9)
  Extended knee: number analyzed (Participants) | 11 | 21 | 26
  Extended knee | -0.4 (0.5) | -0.4 (0.7) | -0.7 (0.9)
  Pes equinovarus: number analyzed (Participants) | 88 | 115 | 120
  Pes equinovarus | -0.7 (0.8) | -0.7 (0.8) | -0.8 (0.8)
  Pes equinovalgus: number analyzed (Participants) | 8 | 10 | 8
  Pes equinovalgus | -0.4 (1.1) | -0.7 (0.7) | -0.3 (0.7)
  Extended hallux: number analyzed (Participants) | 10 | 10 | 19
  Extended hallux | -0.8 (0.9) | -0.9 (1.0) | -0.8 (1.3)
  Flexed toes: number analyzed (Participants) | 27 | 34 | 45
  Flexed toes | -0.5 (0.8) | -0.5 (0.8) | -0.8 (0.7)

7. Secondary Outcome: Change of Ashworth Scale (AS) Score of Every Joint Affected by Clinical Patterns of Spasticity From Study Baseline Visit to Control Visits of Injection Cycles
Description: as for outcome 5
Time Frame: From Study Baseline to Week 4, 16-20 and 28-36
Population: Full analysis set (FAS) - only subjects treated in the respective pattern of respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 155 | 152 | 140
units on a scale
  Internally rotated/extended/adducted shoulder: number analyzed (Participants) | 52 | 68 | 83
  Internally rotated/extended/adducted shoulder | -0.5 (0.8) | -0.6 (0.9) | -0.5 (1.0)
  Flexed elbow: number analyzed (Participants) | 117 | 121 | 122
  Flexed elbow | -0.7 (0.8) | -0.9 (0.8) | -1.2 (0.9)
  Extended elbow: number analyzed (Participants) | 11 | 15 | 19
  Extended elbow | -0.9 (0.8) | -0.7 (0.8) | -0.9 (1.0)
  Pronated forearm: number analyzed (Participants) | 37 | 50 | 47
  Pronated forearm | -1.1 (0.6) | -1.0 (0.9) | -1.1 (0.9)
  Flexed wrist: number analyzed (Participants) | 84 | 85 | 90
  Flexed wrist | -0.9 (0.8) | -1.1 (0.9) | -1.2 (1.1)
  Clenched fist: number analyzed (Participants) | 96 | 108 | 108
  Clenched fist | -0.9 (0.8) | -1.1 (0.9) | -1.4 (0.9)
  Thumb in palm: number analyzed (Participants) | 53 | 61 | 63
  Thumb in palm | -0.9 (1.0) | -1.0 (1.2) | -1.1 (1.3)
  Flexed hip: number analyzed (Participants) | 0 | 0 | 5
  Flexed hip |  |  | -0.6 (1.5)
  Adducted thigh: number analyzed (Participants) | 4 | 7 | 7
  Adducted thigh | -0.3 (0.5) | -0.1 (0.7) | -0.6 (0.8)
  Internally rotated hip: number analyzed (Participants) | 1 | 2 | 3
  Internally rotated hip | -1.0 (NA) — NA = data not available | -0.5 (0.7) | -0.7 (1.5)
  Flexed knee: number analyzed (Participants) | 12 | 23 | 32
  Flexed knee | -0.4 (0.5) | -0.4 (0.8) | -0.4 (1.2)
  Extended knee: number analyzed (Participants) | 11 | 21 | 26
  Extended knee | -0.4 (0.5) | -0.4 (0.6) | -0.6 (0.6)
  Pes equinovarus: number analyzed (Participants) | 88 | 115 | 120
  Pes equinovarus | -0.7 (0.8) | -0.8 (0.9) | -1.1 (0.9)
  Pes equinovalgus: number analyzed (Participants) | 5 | 10 | 8
  Pes equinovalgus | -0.4 (1.1) | -0.9 (0.6) | -0.4 (0.7)
  Extended hallux: number analyzed (Participants) | 10 | 10 | 19
  Extended hallux | -0.8 (0.9) | -0.9 (1.1) | -0.2 (1.3)
  Flexed toes: number analyzed (Participants) | 27 | 34 | 45
  Flexed toes | -0.5 (0.8) | -0.5 (0.7) | -0.6 (0.8)

8. Secondary Outcome: Change of Ashworth Scale (AS) Score of Every Joint Affected by Clinical Patterns of Spasticity From Study Baseline Visit to Injection Cycle Baseline Visits and End of Cycle 3 Visit
Description: as for outcome 5
Time Frame: From Study Baseline to Week 12-16, 24-32 and 36-48
Population: Full analysis set (FAS) - only subjects treated in the respective pattern of respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IncobotulinumtoxinA (Xeomin): Time Frame 1: Time frame 1 is from Study Baseline to Cycle 2 Baseline. Subjects to receive IncobotulinumtoxinA fixed total body dose of 400 units Intramuscular injection.
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 155 | 152 | 140
units on a scale
  Internally rotated/extended/adducted shoulder: number analyzed (Participants) | 69 | 84 | 82
  Internally rotated/extended/adducted shoulder | -0.0 (0.7) | 0.0 (0.9) | -0.3 (0.9)
  Flexed elbow: number analyzed (Participants) | 122 | 124 | 121
  Flexed elbow | -0.2 (0.7) | -0.3 (0.8) | -0.8 (0.9)
  Extended elbow: number analyzed (Participants) | 16 | 19 | 18
  Extended elbow | -0.2 (0.7) | -0.1 (0.9) | -0.2 (0.8)
  Pronated forearm: number analyzed (Participants) | 50 | 48 | 47
  Pronated forearm | -0.3 (0.9) | -0.1 (0.7) | -0.7 (1.0)
  Flexed wrist: number analyzed (Participants) | 87 | 91 | 89
  Flexed wrist | -0.2 (0.7) | -0.2 (1.0) | -0.7 (1.0)
  Clenched fist: number analyzed (Participants) | 110 | 110 | 108
  Clenched fist | -0.2 (0.7) | -0.3 (0.7) | -0.8 (0.9)
  Thumb in palm: number analyzed (Participants) | 63 | 65 | 64
  Thumb in palm | -0.2 (0.9) | -0.3 (0.9) | -0.8 (1.1)
  Flexed hip: number analyzed (Participants) | 0 | 6 | 6
  Flexed hip |  | -0.2 (1.0) | -0.3 (1.4)
  Adducted thigh: number analyzed (Participants) | 7 | 7 | 7
  Adducted thigh | 0 (0) | -0.3 (0.5) | -0.4 (0.8)
  Internally rotated hip: number analyzed (Participants) | 2 | 3 | 3
  Internally rotated hip | -0.5 (0.7) | 0.3 (0.6) | 0.0 (1.0)
  Flexed knee: number analyzed (Participants) | 24 | 32 | 32
  Flexed knee | 0.1 (0.9) | 0.4 (1.2) | -0.4 (1.1)
  Extended knee: number analyzed (Participants) | 22 | 27 | 25
  Extended knee | -0.1 (0.4) | 0.1 (0.5) | -0.4 (0.7)
  Pes equinovarus: number analyzed (Participants) | 117 | 122 | 119
  Pes equinovarus | -0.1 (0.6) | -0.2 (0.7) | -0.7 (0.9)
  Pes equinovalgus: number analyzed (Participants) | 10 | 8 | 7
  Pes equinovalgus | -0.2 (0.4) | -0.1 (0.6) | -0.4 (0.5)
  Extended hallux: number analyzed (Participants) | 10 | 20 | 20
  Extended hallux | 0.0 (1.2) | 0.6 (1.3) | -0.2 (1.0)
  Flexed toes: number analyzed (Participants) | 34 | 45 | 45
  Flexed toes | -0.0 (0.7) | 0.2 (0.7) | -0.4 (0.7)

9. Secondary Outcome: Resistance to Passive Movement Scale (REPAS) Scores of Treated Side
Description: The REPAS is a summary 26-item test used to assess resistance to passive movement in all four limbs of the body. It provides a global evaluation of spasticity status, as well as per hemibody and per limb. 16 items describe the condition of both upper limbs, 10 that of both lower limbs. Each item is rated by using the Ashworth Scale. The sum of the values represent the REPAS score which may range from zero (no resistance for any item) to 104 (limbs rigid for all items). Here, the hemi-REPAS was evaluated, i.e. the maximum value for the treated body side was 52.
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1
Number analyzed (Participants) | 155 | 155 | 152 | 149 | 140 | 138
units on a scale | 24.8 (6.7) | 20.2 (7.1) | 24.0 (7.0) | 18.1 (7.6) | 22.9 (7.2) | 15.7 (7.6)

10. Secondary Outcome: Change of Resistance to Passive Movement Scale (REPAS) Score of Treated Side From Injection Cycle Baseline Visits to Respective Control Visits
Description: as for outcome 9
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 155 | 149 | 138
units on a scale | -4.6 (3.9) | -5.9 (4.2) | -7.1 (4.8)

11. Secondary Outcome: Change of Resistance to Passive Movement Scale (REPAS) Score of Treated Side From Study Baseline Visit to Control Visits of Injection Cycles
Description: as for outcome 9
Time Frame: From Study Baseline to Week 4, 16-20 and 28-36
Population: The full analysis set is the subset of all subjects who were exposed to study medication at least once.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 155 | 149 | 138
units on a scale | -4.6 (3.9) | -6.7 (4.6) | -9.0 (5.5)

12. Secondary Outcome: Change of Resistance to Passive Movement Scale (REPAS) Score of Treated Side From Study Baseline Visit to Injection Cycle Baseline Visits and End of Cycle 3 Visit
Description: as for outcome 9
Time Frame: From Study Baseline to Week 12-16, 24-32 and 36-48
Population: The full analysis set is the subset of all subjects who were exposed to study medication at least once.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IncobotulinumtoxinA (Xeomin): Time Frame1: Time frame 1 is from Study Baseline to Cycle 2 Baseline. Subjects to receive IncobotulinumtoxinA fixed total body dose of 400 units Intramuscular injection.
- IncobotulinumtoxinA (Xeomin): Injection Cycle 3: Time frame 3 is from Study Baseline to End of Cycle 3 Visit. Subjects to receive IncobotulinumtoxinA total body dose of 800 units Intramuscular injection.
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 152 | 140 | 137
units on a scale | -0.8 (4.2) | -1.9 (4.7) | -5.5 (5.3)

13. Secondary Outcome: Functional Ambulation Classification (FAC) Scale Scores
Description: The FAC examines the independence and ambulation of subjects whereby supervision/physical assistance from 1 person is allowed. Subjects are classified to following categories: Level 0: no functional ambulation; Level 1: Ambulator-dependent for physical assistance (Level II); Level 2: Ambulator-dependent for physical assistance (Level I); Level 3: Ambulator-dependent for supervision; Level 4: Ambulator-independent, level surface only; Level 5: Ambulator-independent.
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1
Number analyzed (Participants) | 155 | 155 | 152 | 149 | 140 | 138
units on a scale | 3.5 (1.4) | 3.7 (1.3) | 3.7 (1.3) | 3.8 (1.3) | 3.8 (1.3) | 3.9 (1.2)

14. Secondary Outcome: Change of Functional Ambulation Classification (FAC) Score From Injection Cycle Baseline Visits to Respective Control Visits
Description: as for outcome 13
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 155 | 149 | 138
units on a scale | 0.1 (0.5) | 0.1 (0.4) | 0.1 (0.4)

15. Secondary Outcome: Change of Functional Ambulation Classification (FAC) Score From Study Baseline Visit to Control Visits of Injection Cycles
Description: as for outcome 13
Time Frame: From Study Baseline to Week 4, 16-20 and 28-36
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 155 | 149 | 138
units on a scale | 0.1 (0.5) | 0.3 (0.6) | 0.4 (0.7)

16. Secondary Outcome: Change of Functional Ambulation Classification (FAC) Score From Study Baseline Visit to Injection Cycle Baseline Visits and End of Cycle 3 Visit
Description: as for outcome 13
Time Frame: From Study Baseline to Week 12-16, 24-32 and 36-48
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IncobotulinumtoxinA (Xeomin): Time Frame 1: Time frame 1is from Study Baseline to Cycle 2 Baseline. Subjects to receive IncobotulinumtoxinA fixed total body dose of 400 units Intramuscular injection.
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 152 | 140 | 137
units on a scale | 0.2 (0.5) | 0.3 (0.6) | 0.4 (0.8)

17. Secondary Outcome: Goal Attainment Scale (GAS) Scores for Upper and Lower Limb, Respectively
Description: Change in goal attainment T-scores from respective injection cycle baseline visit. GAS measures the extent to which subject's individual goals are achieved in course of intervention. Subject and treating team have to identify 2 personal goals for each treated limb at each injection cycle. Investigator rates the GAS score for each injection cycle. Degree of goal attainment is rated on 5-point scale (-2, -1, 0, +1, +2; study baseline set to -1) and in order to account for interindividual differences in the number of goals, ratings are computed with the Kiresuk formula (Kiresuk & Sherman, Community Mental Health Journal. 1968;4(6):443-53) resulting in T-scores measuring the degree of goal attainment at each visit. A score of 50 indicates that the individual has reached the expected level of achievement for all goals. The size of change from measurement to measurement indicates incremental change towards or away from goal attainment. Positive values indicate a higher goal attainment.
Time Frame: From Cycle Baseline Visit to Week 12-16, 24-32 and 36-48
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 140 | 138 | 135
units on a scale
  Upper limb | 7.178 (9.254) | 10.601 (9.211) | 13.028 (8.765)
  Lower limb: number analyzed (Participants) | 105 | 126 | 130
  Lower limb | 8.222 (9.649) | 10.914 (9.251) | 13.579 (10.196)

18. Secondary Outcome: Disability Assessment Scale (DAS) Scores in a Selected Principal Therapeutic Target Domain Affecting the Upper Limb
Description: The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which are assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability). One of the domains will be selected per subject per injection cycle. Arithmetic means are built on each patient's target domain value.
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1
Number analyzed (Participants) | 143 | 143 | 151 | 143 | 140 | 128
units on a scale | 2.6 (0.5) | 2.0 (0.7) | 2.4 (0.6) | 1.7 (0.7) | 2.2 (0.6) | 1.5 (0.7)

19. Secondary Outcome: Change of Disability Assessment Scale (DAS) Score in a Selected Principal Therapeutic Target Domain Affecting the Upper Limb From Injection Cycle Baseline Visits to Respective Control Visits
Description: The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which are assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability). One of the domains will be selected per subject per injection cycle. Arithmetic means are built on each patient's target domain value change.
Time Frame: Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 143 | 143 | 128
units on a scale | -0.6 (0.7) | -0.7 (0.7) | -0.7 (0.8)

20. Secondary Outcome: Change of Disability Assessment Scale (DAS) Score in a Selected Principal Therapeutic Target Domain Affecting the Upper Limb From Study Baseline Visit to Control Visits of Injection Cycles
Description: as for outcome 19
Time Frame: From Study Baseline to Week 4, 16-20 and 28-36
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 143 | 143 | 128
units on a scale | -0.6 (0.7) | -0.9 (0.8) | -1.0 (0.9)

21. Primary Outcome: Occurrence of Treatment-Emergent Adverse Events (AEs), AEs of Special Interest (AESIs), and Serious AEs (SAEs) by Injection Cycle, Overall and Related to the Administration of Study Medication
Description: Treatment-emergent Adverse Events (TEASs) are events observed from the time point of first injection until 16 weeks after last injection. Values reported here refer to the number of subjects affected.
Time Frame: From baseline to week 36-48
Population: Safety evaluation set (SES) - only subjects treated in the respective injection cycle were analyzed.
Measure: Number; unit: subjects
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 155 | 152 | 140
subjects
  Any TEAE | 56 | 57 | 36
  Any related TEAE | 7 | 8 | 4
  Any TEAE of special interest | 6 | 8 | 7
  Any related TEAE of special interest | 2 | 4 | 3
  Any serious TEAE | 4 | 11 | 3
  Any related serious TEAE | 0 | 0 | 0

22. Primary Outcome: Investigator's Global Assessment of Tolerability in Subjects
Description: A 4-point Likert scale was used with the ratings 1 = very good, 2 = good, 3 = moderate, and 4 = poor.
Time Frame: Up to Week 48
Population: Safety evaluation set (SES) - only subjects treated in the respective injection cycle were analyzed.
Measure: Number; unit: subjects
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 155 | 152 | 140
subjects
  Very good | 121 | 111 | 117
  Good | 29 | 26 | 20
  Moderate | 3 | 3 | 1
  Poor | 0 | 2 | 0
  Missing | 2 | 10 | 2

23. Secondary Outcome: Change of Disability Assessment Scale (DAS) Score in a Selected Principal Therapeutic Target Domain Affecting the Upper Limb From Study Baseline Visit to Injection Cycle Baseline Visits and End of Cycle 3 Visit.
Description: as for outcome 19
Time Frame: From Study Baseline to Week 12-16, 24-32 and 36-48
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 151 | 140 | 127
units on a scale | -0.2 (0.6) | -0.3 (0.7) | -0.9 (0.9)

24. Secondary Outcome: Global Assessment of Efficacy Scores
Description: Investigator assessment. The global assessment of efficacy will be assessed by the investigator, the subject, and the caregiver using a 4-point Likert scale with the ratings 1 = very good, 2 = good, 3 = moderate, and 4 = poor.
Time Frame: Week 12-16, 24-32 and 36-48
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Number; unit: subjects
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 155 | 152 | 140
subjects
  Frequency 1 (very good) | 7 | 21 | 38
  Frequency 2 (good) | 79 | 89 | 87
  Frequency 3 (moderate) | 63 | 28 | 11
  Frequency 4 (poor) | 3 | 3 | 1
  Missing | 3 | 11 | 3

25. Secondary Outcome: EuroQoL 5-Dimensions Questionnaire (EQ-5D) Scores
Description: The EQ-5D is a common quality of life questionnaire to be filled out by the subject. It evaluates the general impact of a subject's health in 5 dimensions, i.e., on the ability to perform daily physical activities as well as on pain perception and mood. Each dimension is scored on 1 out of 3 categories specific to each dimension, generally meaning: 1= no problem; 2 = moderate problems; 3 = severe problems.
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Number; unit: subjects
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1
Number analyzed (Participants) | 155 | 155 | 152 | 149 | 140 | 138
subjects
  Mobility: Frequency 1 | 12 | 27 | 14 | 24 | 19 | 20
  Mobility: Frequency 2 | 139 | 125 | 136 | 122 | 119 | 116
  Mobility: Frequency 3 | 4 | 3 | 2 | 3 | 2 | 2
  Self-care: Frequency 1: number analyzed (Participants) | 155 | 155 | 152 | 148 | 140 | 138
  Self-care: Frequency 1 | 30 | 31 | 30 | 24 | 24 | 22
  Self-care: Frequency 2: number analyzed (Participants) | 155 | 155 | 152 | 148 | 140 | 138
  Self-care: Frequency 2 | 96 | 100 | 101 | 104 | 101 | 107
  Self-care: Frequency 3: number analyzed (Participants) | 155 | 155 | 152 | 148 | 140 | 138
  Self-care: Frequency 3 | 29 | 24 | 21 | 20 | 15 | 9
  Usual activities: Frequency 1: number analyzed (Participants) | 155 | 155 | 152 | 148 | 140 | 138
  Usual activities: Frequency 1 | 11 | 19 | 16 | 21 | 15 | 17
  Usual activities: Frequency 2 | 113 | 108 | 119 | 110 | 113 | 111
  Usual activities: Frequency 3 | 31 | 28 | 17 | 17 | 12 | 10
  Pain/discomfort: Frequency 1 | 53 | 73 | 56 | 74 | 57 | 77
  Pain/discomfort: Frequency 2 | 85 | 75 | 88 | 70 | 79 | 58
  Pain/discomfort: Frequency 3 | 17 | 7 | 8 | 5 | 4 | 3
  Anxiety/depression: Frequency 1 | 72 | 82 | 83 | 93 | 78 | 85
  Anxiety/depression: Frequency 2 | 69 | 67 | 63 | 49 | 57 | 49
  Anxiety/depression: Frequency 3 | 14 | 6 | 6 | 7 | 5 | 4

26. Secondary Outcome: Visual Analogue Scale (VAS) of EuroQoL 5-Dimensions Questionnaire (EQ-5D) Scores
Description: The EQ-5D is a common quality of life questionnaire to be filled out by the subject. In addition, the subject was to indicate on a visual analogue scale, ranging from 0 to 100, how good or bad their own health was on the examination day (higher values represent better outcome).
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 1 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 2 Control Visit 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3 Baseline Visit | IncobotulinumtoxinA(Xeomin): Injection Cycle 3 Control Visit 1
Number analyzed (Participants) | 154 | 155 | 152 | 149 | 140 | 138
units on a scale | 59.9 (18.9) | 66.7 (17.6) | 67.2 (17.0) | 69.9 (16.6) | 67.1 (17.9) | 68.9 (17.7)

27. Secondary Outcome: Change of EuroQoL 5-dimensions Questionnaire (EQ-5D) Score From Injection Cycle Baseline Visits to Respective Control Visits
Description: The EQ-5D is a common quality of life questionnaire to be filled out by the subject. It evaluates the general impact of a subject's health in 5 dimensions, i.e., on the ability to perform daily physical activities as well as on pain perception and mood. Each dimension is scored on 1 out of 3 categories specific to each dimension, generally meaning: 1= no problem; 2 = moderate problems; 3 = severe problems). In addition, the subject was to indicate on a visual analogue scale, ranging from 0 to 100, how good or bad their own health was on the examination day (higher values indicate better outcome). This table: Frequency -2/-1= improvement by two/one categories; 0 = no change; +1/+2 worsening by one/two categories.
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Number; unit: Subjects
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 155 | 149 | 138
Subjects
  Mobility: Frequency -1 | 18 | 11 | 6
  Mobility: Frequency 0 | 135 | 136 | 128
  Mobility: Frequency 1 | 2 | 2 | 4
  Self-care: Frequency -1: number analyzed (Participants) | 155 | 148 | 138
  Self-care: Frequency -1 | 19 | 7 | 11
  Self-care: Frequency 0: number analyzed (Participants) | 155 | 148 | 138
  Self-care: Frequency 0 | 123 | 127 | 121
  Self-care: Frequency 1: number analyzed (Participants) | 155 | 148 | 138
  Self-care: Frequency 1 | 13 | 14 | 6
  Usual activities: Frequency -2: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency -2 | 0 | 0 | 1
  Usual activities: Frequency -1: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency -1 | 20 | 18 | 7
  Usual activities: Frequency 0: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency 0 | 126 | 116 | 126
  Usual activities: Frequency 1: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency 1 | 9 | 14 | 4
  Pain/discomfort: Frequency -2 | 1 | 2 | 0
  Pain/discomfort: Frequency -1 | 39 | 30 | 29
  Pain/discomfort: Frequency 0 | 105 | 105 | 102
  Pain/discomfort: Frequency 1 | 9 | 12 | 7
  Pain/discomfort: Frequency 2 | 1 | 0 | 0
  Anxiety/depression:Frequency -2 | 0 | 0 | 1
  Anxiety/depression:Frequency -1 | 27 | 18 | 17
  Anxiety/depression: Frequency 0 | 119 | 121 | 111
  Anxiety/depression: Frequency 1 | 9 | 9 | 9
  Anxiety/depression: Frequency 2 | 0 | 1 | 0

28. Secondary Outcome: Change in Visual Analogue Scale of EuroQoL 5-dimensions Questionnaire (EQ-5D) Score From Injection Cycle Baseline Visits to Respective Control Visits
Description: as for outcome 26
Time Frame: From Cycle Baseline to Week 4 of Each Cycle
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 154 | 149 | 138
units on a scale | 6.7 (14.1) | 2.4 (12.4) | 1.7 (12.4)

29. Secondary Outcome: Change of EuroQoL 5-dimensions Questionnaire (EQ-5D) Score From Study Baseline Visit to Control Visits of Injection Cycles
Description: as for outcome 27
Time Frame: From Study Baseline to Week 4, 16-20 and 28-36
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Number; unit: subjects
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 155 | 149 | 138
subjects
  Mobility: Frequency -1 | 18 | 16 | 14
  Mobility: Frequency 0 | 135 | 127 | 118
  Mobility: Frequency 1 | 2 | 5 | 5
  Self-care: Frequency -1: number analyzed (Participants) | 155 | 148 | 138
  Self-care: Frequency -1 | 19 | 20 | 25
  Self-care: Frequency 0: number analyzed (Participants) | 155 | 148 | 138
  Self-care: Frequency 0 | 123 | 110 | 100
  Self-care: Frequency 1: number analyzed (Participants) | 155 | 148 | 138
  Self-care: Frequency 1 | 13 | 18 | 13
  Usual activities: Frequency -2: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency -2 | 0 | 1 | 1
  Usual activities: Frequency -1: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency -1 | 20 | 31 | 31
  Usual activities: Frequency 0: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency 0 | 126 | 103 | 98
  Usual activities: Frequency 1: number analyzed (Participants) | 155 | 148 | 138
  Usual activities: Frequency 1 | 9 | 13 | 8
  Pain/discomfort: Frequency -2 | 1 | 3 | 3
  Pain/discomfort: Frequency -1 | 39 | 40 | 42
  Pain/discomfort: Frequency 0 | 105 | 93 | 85
  Pain/discomfort: Frequency 1 | 9 | 13 | 8
  Pain/discomfort: Frequency 2 | 1 | 0 | 0
  Anxiety/depression:Frequency -2 | 0 | 7 | 6
  Anxiety/depression:Frequency -1 | 27 | 28 | 32
  Anxiety/depression:Frequency 0 | 119 | 100 | 85
  Anxiety/depression:Frequency 1 | 9 | 14 | 15
  Anxiety/depression:Frequency 2 | 0 | 0 | 0

30. Secondary Outcome: Change in Visual Analogue Scale of EuroQoL 5-dimensions Questionnaire (EQ-5D) Score From Study Baseline Visit to Control Visits of Injection Cycles
Description: The EQ-5D is a common quality of life questionnaire to be filled out by the subject. It evaluates the general impact of a subject's health in 5 dimensions, i.e., on the ability to perform daily physical activities as well as on pain perception and mood. Each dimension is scored on 1 out of 3 categories specific to each dimension, generally meaning: 1= no problem; 2 = moderate problems; 3 = severe problems). In addition, the subject was to indicate on a visual analogue scale, ranging from 0 to 100, how good or bad their own health was on the examination day (higher values indicate better outcome). This table: Positive values indicate improvement
Time Frame: From Study Baseline to Week 4, 16-20 and 28-36
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Injection Cycle 1 | IncobotulinumtoxinA (Xeomin): Injection Cycle 2 | IncobotulinumtoxinA (Xeomin): Injection Cycle 3
Number analyzed (Participants) | 154 | 148 | 137
units on a scale | 6.7 (14.1) | 9.6 (16.3) | 8.6 (17.0)

31. Secondary Outcome: Change of EuroQoL 5-dimensions Questionnaire (EQ-5D) Score From Study Baseline Visit to Injection Cycle Baseline Visits and End of Cycle 3 Visit
Description: as for outcome 27
Time Frame: From Study Baseline to Week 12-16, 24-32 and 36-48
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Number; unit: subjects
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 152 | 140 | 137
subjects
  Mobility: Frequency -1 | 10 | 13 | 16
  Mobility: Frequency 0 | 137 | 121 | 116
  Mobility: Frequency 1 | 5 | 5 | 4
  Self-care: Frequency -1 | 20 | 24 | 30
  Self-care: Frequency 0 | 120 | 99 | 97
  Self-care: Frequency 1 | 12 | 17 | 10
  Usual activities: Frequency -2 | 1 | 1 | 1
  Usual activities: Frequency -1 | 21 | 26 | 33
  Usual activities: Frequency 0 | 125 | 106 | 96
  Usual activities: Frequency 1 | 5 | 7 | 7
  Pain/discomfort: Frequency -2 | 0 | 0 | 3
  Pain/discomfort: Frequency -1 | 32 | 35 | 40
  Pain/discomfort: Frequency 0 | 100 | 89 | 81
  Pain/discomfort: Frequency 1 | 20 | 15 | 13
  Pain/discomfort: Frequency 2 | 0 | 1 | 0
  Anxiety/depression: Frequency -2 | 2 | 4 | 5
  Anxiety/depression: Frequency -1 | 29 | 28 | 30
  Anxiety/depression: Frequency 0 | 108 | 91 | 89
  Anxiety/depression: Frequency 1 | 12 | 17 | 13
  Anxiety/depression: Frequency 2 | 1 | 0 | 0

32. Secondary Outcome: Change in Visual Analogue Scale of EuroQoL 5-dimensions Questionnaire (EQ-5D) Score From Study Baseline Visit to Injection Cycle Baseline Visits and End of Cycle 3 Visit
Description: as for outcome 30
Time Frame: From Study Baseline to Week 12-16, 24-32 and 36-48
Population: Full analysis set (FAS) - only subjects treated in the respective injection cycle were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IncobotulinumtoxinA (Xeomin): Time Frame 1 | IncobotulinumtoxinA (Xeomin): Time Frame 2 | IncobotulinumtoxinA (Xeomin): Time Frame 3
Number analyzed (Participants) | 151 | 139 | 136
units on a scale | 7.1 (16.3) | 6.9 (15.8) | 10.5 (17.5)

ADVERSE EVENTS:
Time Frame: From the time point of first injection until 16 weeks after last injection
Arm/Group | IncobotulinumtoxinA (Xeomin) (up to 800 Units)
Serious Adverse Events (participants affected / at risk) | 17/155
Other Adverse Events (participants affected / at risk) | 34/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IncobotulinumtoxinA (Xeomin) (up to 800 Units) (N=155)
Convulsion (Nervous system disorders) | 4
Epilepsy (Nervous system disorders) | 3
Cerebral infarction (Nervous system disorders) | 2
Ischemic stroke (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Meningitis bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Cardiac failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IncobotulinumtoxinA (Xeomin) (up to 800 Units) (N=155)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 12 (17)
Diarrhoea (Gastrointestinal disorders) | 10 (13)
Nasopharyngitis (Infections and infestations) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the Investigator will consider these doubts in the publication as long as the scientific neutrality is not affected.